CLINICAL TRIAL: NCT01580592
Title: A Two-center, Double Blind, Placebo-controlled Study in Parallel Design to Assess the Efficacy and Safety of 150 and 300 mg Omalizumab in Subjects With Antihistamine-resistant Cold Contact Urticaria (CCU)
Brief Title: Cold Urticaria Treatment With Xolair
Acronym: CUTEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Martin Metz, Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIGE025EDE14T
Record Dates: First submitted 2012-04-18; First posted 2012-04-19 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Cold Contact Urticaria
MeSH Terms: conditions — Cold Urticaria | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Omalizumab 150mg (Experimental)
  Interventions: Drug: Omalizumab
- Omalizumab 300mg (Experimental)
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — 150mg, s.c., every 4 weeks
  Other Names: Xolair
  Arms: Omalizumab 150mg
Drug: Omalizumab — 300mg, s.c., every 4 weeks
  Other Names: Xolair
  Arms: Omalizumab 300mg
Drug: Placebo — Placebo, s.c., every 4 weeks
  Arms: Placebo

SUMMARY:
Urticaria is a very frequent skin condition characterised by transient wheal and flare type skin reactions associated with severe pruritus. Cold contact urticaria (CCU) is a frequent form of physical urticaria that is characterized by the development of wheal and flare type skin reactions due to the release of histamine and other proinflammatory mast cell mediators following exposure of the skin to cold. Among all physical urticaria subtypes the frequency of CCU varies between 5.7% and 33.8% in different studies. Physical urticarias including CCU are known to severely impair the quality of life of affected patients.

The treatment of choice in CCU, as well as in other inducible forms and spontaneous urticaria, are non-sedating H1 antihistamines. Recent data have shown that updosing of H1 blockers is significantly more effective in reducing symptoms in cold urticaria than standard-dose treatment. Thus, patients who cannot be sufficiently controlled with standard-dose antihistamines should receive high-dose H1 blockers up to 4 times the standard dose as recommended by the new international guidelines for the management of urticaria.

Previous phase II studies in patients with chronic spontaneous urticaria have shown favorable results for the treatment with omalizumab (Xolair®). Proof-of-concept data from completed studies suggest that omalizumab improves urticaria in patients with chronic spontaneous urticaria who have failed treatment with H1 antihistamines as well as those who have failed treatment with a combination of H1 and H2 antihistamines and a leukotriene receptor antagonist. In addition, two case reports of patients with severe therapy refractory CCU treated with omalizumab reported a complete response with no urticarial symptoms after cold challenge. In summary, these data suggest that omalizumab may have a beneficial effect in the treatment of CCU.

ELIGIBILITY:
Inclusion Criteria:

Adults (18 years or older) Informed consent signed and dated Able to read, understand and willing to sign the informed consent form and abide with study procedures Diagnosis of CCU lasting for at least 6 months Willing, committed and able to return for all clinic visits and complete all study-related procedures, including willingness to have SC injections administered by a qualified person In females of childbearing potential: Negative pregnancy test; females willing to use highly effective contraception (Pearl-Index < 1). A woman will be considered not of childbearing potential if she is post-menopausal for greater than two years or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) No participation in other clinical trials 4 weeks before and after participation in this study

Exclusion Criteria:

Patients with acute urticaria Concurrent/ongoing treatment with immunosuppressives (e.g. systemic steroids, cyclosporine, methotrexate, dapsone or others) within 4 weeks or 5 half lives prior to day 0, whichever is longer Significant medical condition rendering the patient immunocompromised or not suitable for a clinical trial Significant concomitant illness that would adversely affect the subject's participation or evaluation in this study History of malignancies within five years prior to screening other than a successfully treated non-metastatic cutaneous, basal, or squamous cell carcinoma and/or in situ cancer Presence of clinically significant laboratory abnormalities Lactating females or pregnant females Subjects for whom there is concern about compliance with the protocol procedures Any medical condition which, in the opinion of the Investigator, would interfere with participation in the study or place the subject at risk History of substance abuse (drug or alcohol) or any other factor (e.g., serious psychiatric condition) within the last 5 years that could limit the subject's ability to comply with study procedures Subjects who are detained officially or legally to an official institute Previous use of omalizumab within the last 6 months Intake of antihistamines or leukotriene antagonists within 7 days prior to visit 1 Intake of oral corticosteroids within 14 days prior to visit 1 Use of depot corticosteroids or chronic systemic corticosteroids within 21 days before beginning of the study Known hypersensitivity to any ingredients, including excipients (sucrose, histidine, polysorbate 20) of the study medication or drugs related to omalizumab (e.g.: monoclonal antibodies, polyclonal gammaglobulin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Metz, MD, Principal Investigator — Charité
Locations (3):
- Germany (3):
  - University Aachen, Aachen
  - Allergie-Centrum-Charité, Charité - Universitätsmedizin Berlin, Berlin
  - Hautklinik Mainz, Mainz

REFERENCES:
- [Derived] Metz M, Schutz A, Weller K, Gorczyza M, Zimmer S, Staubach P, Merk HF, Maurer M. Omalizumab is effective in cold urticaria-results of a randomized placebo-controlled trial. J Allergy Clin Immunol. 2017 Sep;140(3):864-867.e5. doi: 10.1016/j.jaci.2017.01.043. Epub 2017 Apr 4. No abstract available. PMID 28389393

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo
Started | 10 | 9 | 12
Completed | 10 | 9 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 12 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 12 | 31
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 9 | 23
  Male | 3 | 2 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 9 | 12 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 10 | 9 | 12 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Critical Temperature Thresholds (CTT) From Baseline to Day 70 After Treatment With Omalizumab Compared to Placebo
Description: The primary efficacy outcome was the change in trigger thresholds from baseline to week ten using TempTest® to assess critical temperature thresholds in °C.
Time Frame: day 70
Population: female and male
Measure: Mean (Standard Deviation); unit: degree celcius
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo
Number analyzed (Participants) | 10 | 9 | 12
degree celcius | -10.6 (7.6) | -10.4 (9.4) | -0.3 (3.9)
Statistical Analysis 1: Comparison: Omalizumab 150mg; Test type: Superiority or Other; p = 0.001, ANOVA; Mean Difference (Final Values) = -10.6, Standard Deviation 7.6 — for omalizumab 150mg
Statistical Analysis 2: Comparison: Omalizumab 300mg; Test type: Superiority or Other; p = 0.01, ANOVA; Mean Difference (Final Values) = 10.4, Standard Deviation 9.4
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.3, Standard Deviation 3.9

2. Secondary Outcome: Number of Participants With Abnormal Physical Examinations, Laboratory Assessments, Vital Signs, and Adverse Events
Description: This includes physical examination, routine safety laboratory assessments, vital signs and adverse event reporting
Time Frame: day 70
Measure: Number; unit: participants
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo
Number analyzed (Participants) | 10 | 9 | 12
participants | 7 | 7 | 9
Statistical Analysis 1: Comparison: Omalizumab 150mg vs Omalizumab 300mg vs Placebo; Test type: Superiority or Other; p = 0.988, Chi-squared

ADVERSE EVENTS:
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 4/10 | 4/9 | 5/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab 150mg (N=10) | Omalizumab 300mg (N=9) | Placebo (N=12)
Headache (General disorders) | 2 | 2 | 4
upper respiratory tract infection (Infections and infestations) | 2 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No